CLINICAL TRIAL: NCT06526104
Title: Phase II Single Arm Study of Tremelimumab and Durvalumab (MEDI4736) (T300+D) in Advanced Hepatocellular Carcinomas With Child-Pugh-B Cirrhosis (STRIDE in CP-B)
Brief Title: Study of Tremelimumab and Durvalumab (MEDI4736) (T300+D) in Advanced Hepatocellular Carcinomas With Child-Pugh-B Cirrhosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sukeshi Patel, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 23-0164; STUDY00001088 (Other: University of Texas Health Science Center at San Antonio)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis, Liver
Keywords: Tremelimumab; Durvalumab; Child-Pugh-B Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm, phase II study of patients with advanced HCC with Child-Pugh B cirrhosis who are eligible for first-line treatment with T300+D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stride (Single T Regular Interval D) Arm (Experimental): Tremelimumab dosed once at the beginning of the first cycle, 300mg IV infusion and Durvalumab 1500mg IV dosed with the first dose of Tremelimumab and then once per cycle (every 4 weeks)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tremelimumab — Priming dose of tremelimumab 300 mg IV once (Cycle 1, Day 1 only)
  Other Names: Imjudo
Drug: Durvalumab — Durvalumab 1500 mg IV on Day 1 of each 4-week cycle.
  Other Names: Imfinzi

SUMMARY:
This is a single-arm, phase II study of patients with advanced liver cancer or hepatocellular carcinoma (HCC) who are eligible for first-line treatment with T300+D. The invesitgators hypothesize that T300+D will be safe and tolerated in CP-B patients with HCC. HCC mostly affects disadvantaged populations with higher rates among racial/ethnic minorities, who are often not included in clinical trials (i.e., Hispanics, Blacks, underserved, low socioeconomic status) and present with more severe disease. Given there is not much data in the US patient cohort, this study provides a chance to gain that knowledge.

DETAILED DESCRIPTION:
Priming dose of tremelimumab 300 mg IV once (Cycle 1, Day 1 only) with durvalumab 1500 mg IV on Day 1 of each 4-week cycle. Patients will stay on study treatment until evidence of disease progression, unacceptable toxicity, or death.

All eligible patients who consent to this study must have a baseline evaluation (CT or MRI) within 28 days of the start of treatment.

Follow-up: A repeat CT/MRI scan will be performed after 2 cycles of treatment regimen to evaluate response based on RECIST 1.1 criteria (See Appendix for definitions of response).12 Serum tumor marker AFP (every cycle) and CT/MRI scans will be repeated at least every 2 cycles, or 8 weeks, to ensure no progression of disease. Patients will continue treatment until disease progression, unacceptable toxicity, withdrawal of consent by the patient, or decision of physician for patient's best interest. Each patient will be followed for survival for up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with HCC based on pathologic diagnosis from biopsy or radiographic diagnosis on CT liver or MRI liver (i.e., Barcelona Clinic Liver Cancer (BCLC) stage B and not candidate for locoregional therapies or BCLC stage C)10
2. Patients with Child-Pugh-B7 or -B8 liver cirrhosis11
3. ECOG performance status score 0-1
4. Patients with Hepatitis B Virus (HBV) infection are required to receive effective antiviral therapy and have a viral load less than 500 IU/mL at screening; antiviral therapy is not required for patients with Hepatitis C Virus (HCV) infection.
5. Adequate organ and bone marrow function:

   1. Absolute neutrophil counts ≥1000/uL
   2. Platelets ≥60 × 100/uL
   3. Hemoglobin ≥8.0 g/dL
   4. ALT and AST ≤5× upper limit of normal each
   5. Bilirubin ≤3 mg/dL,
   6. International normalized ratio (INR) ≤2.3 or prothrombin time ≤6 seconds above control)
   7. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min)=Weight (kg) x (140 - Age) /72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min)=Weight (kg) x (140 - Age) x 0.85 /72 x serum creatinine (mg/dL)
6. Body weight >30 kilogram (kg)
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
8. Age >18 years at time of study entry or adult male or female (according to age of majority as defined as ≥18 years)
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. Must have a life expectancy of at least 12 weeks.
11. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline.

Exclusion Criteria:

1. Patients who are candidates for curative treatments
2. History of uncontrolled hepatic encephalopathy in the past 6 months; patients who are stable on medical therapy are eligible.
3. Active substance abuse or alcohol abuse at the time of consent or enrollment, which in the opinion of the treating physician would interfere with the safety of the patient and/or adherence to the study protocol.
4. Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
5. Prior systemic therapy for locally advanced or metastatic HCC
6. Participation in another clinical study with an investigational product during the last 1 month.
7. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
8. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable. <<amend as required based on any combination studies with other anticancer agents>>
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
11. History of allogenic organ transplantation
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
    5. Patients with celiac disease controlled by diet alone.
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
14. History of leptomeningeal carcinomatosis
15. History of active primary immunodeficiency
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab and tremelimumab combination therapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
21. Known allergy or hypersensitivity to IP or any excipient.
22. History of another primary malignancy except for:

    1. Malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk for recurrence.
    2. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or lentigo maligna that has undergone potentially curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or Higher Treatment Related Treatment Emergent-Adverse Events (TRTE-AEs) | Baseline up to 1 year
  The number and grade 1-5 of all adverse events will be documented according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0; measured at baseline, each cycle, and up to 90 days after treatment discontinued. Grade 3 and higher TRTE-AEs will be reported for this outcome.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to 1 year
  ORR, complete and partial response, confirmed and unconfirmed as defined by Response evaluation criteria in solid tumors (RECIST) v1.1.9. ORR, complete and partial response, confirmed and unconfirmed) as defined by RECIST v1.1.9. RECIST version 1.1 RECIST is used as tumor response criteria in most trials of solid tumors in general. RECIST1. 1 uses unidimensional diameters of target lesions and the sum of measurements of all target lesions as a quantitative measure of tumor burden.
Progression Free Survival (PFS) | Baseline to 1 year
  Measured from the date of registration until disease progression, symptomatic deterioration, or death.
Overall Survival (OS) | Baseline to 1 year
  Measured from date of registration until death
Albumin-Bilirubin (ALBI) grade | Baseline to 1 year
  Albumin-bilirubin (ALBI) grade is a tool that assesses liver function by combining serum albumin and bilirubin levels. It can be used to predict the prognosis of patients with liver cirrhosis and hepatocellular carcinoma, and has been shown to be more accurate than the Child-Pugh score. ALBI grade can also be used to predict survival for patients treated with radioembolization (RE), and as a prognostic indicator for cancer patients receiving chemotherapy. A calculator is used to generate the score. Based on the score, patients are graded between grade 1 (lowest mortality risk, ALBI score ≤2.60) and grade 3 the highest mortality risk (score >-1.39).

OTHER OUTCOMES:
European Organisation For Research and Treatment of Cancer (EORTC)- Quality of Life Questionnaire (QLC) | Baseline up to 16 weeks
  A 30-item self-administered questionnaire with 9 multiple-item scales: 5 scales that assess aspects of functioning (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), and a global measure of health status/QOL scale. There are 5 single-item measures assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and 1 item concerning the perceived financial impact of the disease. All but 2 questions have 4-point scales: "Not at all," "A little," "Quite a bit," and "Very much". The 2 questions concerning global health status and QOL have 7-point scales with ratings ranging from "Very poor" to "Excellent". For each of the 15 domains (9 multiple item scales and 6 single-item scales), final scores are transformed such that they range from 0 to 100, where higher scores indicate greater functioning, greater health related quality of life, or lower level of symptoms.
EORTC QLQ-HCC18 (18-item hepatocellular cancer health-related quality of life questionnaire) | Baseline to 16 weeks
  The EORTC QLQ-HCC18 module is an 18-item self-administered questionnaire (Appendix) developed and validated specifically for HCC). There are 5 multiple-item symptom scales (fatigue [3 items], jaundice [2 items], nutrition [5 items], pain [2 items], and fever [2 items]); 2 single-item symptom scales (abdominal swelling and sexual interest); and 1 multiple-item functional scale (body image [2 items]). All questions have a 4-point scale: "Not at all," "A little," "Quite a bit," and "Very much". For each of the 8 domains (6 multiple-item scales and 2 single-item scales), final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms. All item response scores are converted into 0 to 100 scores; for all scales, a higher score means a worse symptom or a poorer health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Arora, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Any manuscript, abstract or other publication or presentation of results or information arising in connection with the trial (including any ancillary trial involving trial subjects) must be prepared in conjunction with the Mays DSMB, the trial's statistician, and verification that all study data to be used for the publication has been monitored for accuracy by the Mays QA team prior to publication or presentation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the completion of the study at the time of publication in a peer review journal.